CLINICAL TRIAL: NCT04902235
Title: Identification and Clinical Relevance of an Oxytocin Deficient State: a Randomized, Crossover, Placebo-controlled, Proof-of-concept Physiopathological Study (CRH Study)
Brief Title: Identification and Clinical Relevance of an Oxytocin Deficient State (CRH Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: IIBSP-OXI-2020-101
Record Dates: First submitted 2021-05-17; First posted 2021-05-26 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2022-03

CONDITIONS: Hypopituitarism; Central Diabetes Insipidus; Panhypopituitarism; Psychological Disorder; Social Isolation; Hypothalamic Diseases; Pituitary Diseases; Oxytocin Deficiency
Keywords: oxytocin; panhypopituitarism; central diabetes insipidus; hypothalamus-pituitary diseases; cortisol; ACTH; corticorelin hormone
MeSH Terms: conditions — Hypopituitarism; Diabetes Insipidus, Neurogenic; Combined Pituitary Hormone Deficiency; Mental Disorders; Social Isolation; Hypothalamic Diseases; Pituitary Diseases

STUDY DESIGN:
Intervention Model Description: Single-blind, randomized, placebo-controlled proof-of-concept studies with a crossover assignment
Who Masked: Participant
Masking Description: participants will be blinded to the intervention assignment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CRH administration (Experimental): Experimental: CRH administration
  Interventions: Drug: Experimental: CRH administration
- Placebo administration (Placebo Comparator): Control: Placebo administration
  Interventions: Drug: Control: Placebo administration

INTERVENTIONS:
Drug: Experimental: CRH administration — CRH at 1.0 µg/kg/body weight will be injected intravenously as a bolus over 30 seconds and samples will be collected over 2 hours (15 (T15), 30 (T30), 45 (T45), 60 (T60'), 90 (T90) and 120 (T120) minutes) after CRH:placebo administration to assess OT secretory patterns
  Arms: CRH administration
Drug: Control: Placebo administration — Sodium Chloride 0.9% will be administered intravenously as a bolus over 30 seconds at equivalent volume than CRH administration (1.0 µg/kg/body weight)
  Arms: Placebo administration

SUMMARY:
Oxytocin (OT) is a hypothalamic peptide that enters the peripheral circulation via the posterior pituitary gland. OT plays a key role in regulating appetite, psychopathology, prosocial behavior and sexual function. Hypopituitarism is associated with increased obesity, increased psychopathology, sexual and prosocial dysfunction despite appropriate hormone replacement. A few studies suggest the existence of a possible OT deficient state in hypopituitarism. In animal models, corticorelin hormone (CRH) has shown to increase OT release.

This study is designed to evaluate oxytocin values after administration of CRH in adults (healthy volunteers and patients with hypopituitarism).

The investigators hypothesize that OT response will be blunted following CRH in patients with hypopituitarism compared to healthy controls.

DETAILED DESCRIPTION:
This research is focused on two groups of participants: healthy controls (HC) and hypopituitary patients (HYPO) with at least one symptom of hypothalamic damage, presumably at highest risk for OT deficiency.

The aim is to improve knowledge on the physiology and patho-physiology of endogenous OT secretion in hypopituitary patients compared to healthy controls using a randomized, single-blind, crossover assignment (CRH vs placebo), placebo-control design.

Clinical implications of secretory OT dynamics and release under different stimuli using validated questionnaires to evaluate psychopathology, socio-emotional functioning, disordered eating behavior, impaired quality of life and sexual dysfunction, will be also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hypopituitarism (HYPO) (>1 pituitary hormone deficiency) and stable hormone replacement for the prior three months
* At least one clinical sign of hypothalamic damage
* Female participants will be done in the early to midfollicular phase

Exclusion Criteria:

* uncorrected hormone deficiency
* creatinine >1.5mg/dL
* alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2.5x upper limit of normal
* hematocrit less than 30%
* suicidality or active psychosis
* participation in a trial with investigational drugs within 30 days
* using a high glucocorticoid dose
* vigorous physical exercise
* alcohol intake within 24 hours before the study participation
* evidence of any acute illness or any illness that the Investigator determines could interfere with study participation or safety
* pregnancy or breastfeeding for last 8 weeks
* known allergies towards CRH
* patients refusing or unable to give written informed consent
* Additionally for healthy controls: the presence of brain or pituitary tumor, radiation involving the hypothalamus or pituitary, history of hypopituitarism or receiving testosterone or glucocorticoids esters.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Change in oxytocin concentration | Baseline blood exam (timepoint 0) and further blood collections after 15, 30, 45, 60, 90 and 120 minutes after baseline blood collection
  Change in oxytocin concentration (pg/mL) after administration of 1.0 µg/kg/body weight of CRH or 0.9% sodium chloride (NaCl)

SECONDARY OUTCOMES:
Maximal change in oxytocin concentration (pg/mL) | Within the two hours after the injection
  Maximal change in oxytocin concentration (pg/mL) after administration of 1.0 µg/kg/body weight of CRH or 0.9% NaCl
Overall oxytocin secretion | Within the two hours after the injection
  Oxytocin area under the curve after administration of 1.0 µg/kg/body weight of CRH or 0.9% NaCl
Change in cortisol concentration (nmol/L) | Baseline blood exam (timepoint 0) and further blood collections after 15, 30, 45, 60, 90 and 120 minutes after baseline blood collection
  Change in cortisol concentration (nmol/L) after administration of 1.0 µg/kg/body weight of CRH or 0.9% NaCl
Change in adrenocorticotropic hormone (ACTH) values | Baseline blood exam (timepoint 0) and further blood collections after 15, 30, 45, 60, 90 and 120 minutes after baseline blood collection
  Change in ACTH values (pmol/L) after administration of 1.0 µg/kg/body weight of CRH or 0.9% NaCl
Mood assessment | Baseline
  Correlation between Beck Depression Inventory-2 score (range from 0 to 63, higher scores mean a worse outcome) and baseline oxytocin concentration (pg/mL)
Quality of life assessment | Baseline
  Correlation between 36 item- Short Form Health Survey score (range from 0 to 100, the higher scores indicate better health status) and baseline oxytocin concentration (pg/mL)
Impulsivity assessment | Baseline
  Correlation between Barratt Impulsiveness Scale (range from 30 to 120, higher scores indicate greater impulsivity) and baseline oxytocin concentration (pg/mL)
Alexithymia assessment | Baseline
  Correlation between Toronto Alexithymia scales-20 score (range from 20 to 100, higher scores mean a worse outcome) and baseline oxytocin concentration (pg/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Aulinas, MD PhD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

REFERENCES:
- [Derived] Asla Q, Garrido M, Urgell E, Terzan S, Santos A, Fernandez M, Varghese N, Atila C, Calabrese A, Biagetti B, Plessow F, Gich I, Christ-Crain M, Eckert A, Webb SM, Lawson EA, Aulinas A. Oxytocin levels in response to CRH administration in hypopituitarism and hypothalamic damage: a randomized, crossover, placebo-controlled trial. Sci Rep. 2025 Jan 18;15(1):2360. doi: 10.1038/s41598-025-86566-y. PMID 39824923